CLINICAL TRIAL: NCT01757691
Title: A 48-week, Double-blind, Randomized, Multi-center, Parallel-group Study Comparing Structural Changes in the Retina and Evolution of Visual Function After Immediate Versus Delayed Treatment With Fingolimod in Patients With Acute Demyelinating Optic Neuritis
Brief Title: Fingolimod (FTY720) in Acute Demyelinating Optic Neuritis (ADON)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of this study was based on Novartis decision to discontinue development of fingolimod for the treatment of ADON
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D2402; 2012-002968-27 (EudraCT Number)
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Acute Demylelinating Optic Neuritis
Keywords: Acute demyelinating optic neuritis; Optic neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fingolimod 0.5mg/daily (Experimental): Oral capsule dose was given once daily for 48 weeks
  Interventions: Drug: Fingolimod 0.5mg/daily
- Placebo (Placebo Comparator): Patients received oral dose of placebo from Weeks 0-18, followed by oral dose of fingolimod 0.5/mg capsule from Weeks 18-48
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fingolimod 0.5mg/daily
  Other Names: FTY, Gilenya
  Arms: Fingolimod 0.5mg/daily
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of fingolimod 0.5mg versus placebo in patients with suspected acute demyelinating optic neuritis (ADON) receiving standard steroid treatment

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms of ADON in one eye (loss of vision, pain on movement, impairment of color vision)
* First episode of ADON
* Able to undergo treatment with IV steroids

Exclusion Criteria:

* History of any unexplained eye or neurological symptoms lasting longer than 48 hours
* Optic neuritis in both eyes
* Concomitant condition in either eye, other than optic neuritis
* History of heart condition/disease
* Patients with uncontrolled diabetes mellitus
* Patients with liver conditions/disease
* Inability to undergo MRI
* Pregnant or nursing women
* Women of childbearing potential who are not using highly effective method of birth control

  * Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, St. Petersburg, Florida, United States
- Novartis Investigative Site, Majadahonda, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fingolimod 0.5mg/Daily | Placebo
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Administrative problems | 2 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fingolimod 0.5mg/Daily
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Retinal Nerve Fiber Layer (RNFL) Thinning in Patients Treated With Fingolimod 0.5mg/Day, Relative to Patients Treated With Placebo
Description: Due to early termination and low patient enrollment the primary outcome measure was not analyzed
Time Frame: Baseline and Week 18
Arm/Group | Fingolimod 0.5mg/Daily | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Low Contrast Visual Acuity (LCVA)
Description: Due to early termination and low patient enrollment this trial was not powered for efficacy
Time Frame: Baseline, Week 48
Arm/Group | Fingolimod 0.5mg/Daily | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Vision Based Quality of Life (QoL) Utility Score
Description: Due to early termination and low patient enrollment this trial was not powered for efficacy
Time Frame: Baseline, Week 18, Week 48
Arm/Group | Fingolimod 0.5mg/Daily | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Paatients Converting to Either 2005 or 2010 McDonald MS or to CDMS
Description: Due to early termination and low patient enrollment this trial was not powered for efficacy
Time Frame: Baseline, Week 18, Week 48
Arm/Group | Fingolimod 0.5mg/Daily | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Particpants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of particpants with Adverse events as a measure of safety and tolerability
Time Frame: Weeks 0, 4, 8, 12, 18, 24, 36, 48, 60
Population: Safety population consited of all patients who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Fingolimod 0.5mg/Daily
Number analyzed (Participants) | 2
Participants
  Adverse Events (AE) | 1
  Death | 0
  Non -Fatal Seriuos Aderse Event (SAE) | 0

ADVERSE EVENTS:
Description: Safety population consited of all patients who received at least one dose of study medication
Arm/Group | Fingolimod 0.5mg/Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5mg/Daily (N=2) | Placebo (N=0)
Vomiting (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
ASTHMA EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis doesn not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e. data from all sites) in the clinical trial or disclosure of the trial results in their entirety.